CLINICAL TRIAL: NCT07255820
Title: Comparative Efficacy and Safety of Dual Versus Triple Lipid-Lowering Therapies (Rosuvastatin/Ezetimibe, Bempedoic Acid/Ezetimibe, and Rosuvastatin/Ezetimibe/Bempedoic Acid ) in Type 2 Diabetes Mellitus Patients With Elevated LDL Cholesterol
Brief Title: Dual vs Triple Lipid-Lowering Therapy in Type 2 Diabetes Mellitus Patients With Elevated LDL Cholesterol
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUHS-IRB # 180/25
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus; Hypercholesterolemia / Elevated LDL Cholesterol
Keywords: Lipid-lowering therapy,; Rosuvastatin, Ezetimibe, Bempedoic Acid; Dual therapy vs Triple therapy; LDL-C; Dyslipidemia; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia; Hyperlipoproteinemia Type II; Dyslipidemias | interventions — Rosuvastatin Calcium; Ezetimibe; 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rosuvastatin + Ezetimibe (Active Comparator): Rosuvastatin is a statin that lowers LDL cholesterol by inhibiting HMG-CoA reductase. Ezetimibe inhibits cholesterol absorption in the intestine.
  Interventions: Drug: Rosuvastatin + Ezetimibe
- Bempedoic Acid + Ezetimibe (Active Comparator): Bempedoic acid is an ATP citrate lyase inhibitor that reduces LDL cholesterol. Ezetimibe inhibits diatery cholesterol absorption in the intestine
  Interventions: Drug: Bempedoic Acid + Ezetimibe
- Rosuvastatin + Ezetimibe + Bempedoic Acid (Active Comparator): This triple therapy combines statin therapy with cholesterol absorption inhibition and ATP citrate lyase inhibition to optimize LDL reduction.
  Interventions: Drug: Rosuvastatin + Ezetimibe + Bempedoic Acid

INTERVENTIONS:
Drug: Rosuvastatin + Ezetimibe — Group A (Dual therapy 1): Tab Rosuvastatin 20 mg + Tab Ezetimibe 10mg (FDC) orally, once daily for 90 days
  Arms: Rosuvastatin + Ezetimibe
Drug: Bempedoic Acid + Ezetimibe — Group B (Dual therapy 2): Tab Bempedoic Acid 180mg+ Tab Ezetimibe 10mg (FDC) orally, once daily for 90 days
  Arms: Bempedoic Acid + Ezetimibe
Drug: Rosuvastatin + Ezetimibe + Bempedoic Acid — Group C (Triple therapy): Tab Rosuvastatin 20 mg+ Tab Ezetimibe 10mg+ Tab Bempedoic Acid 180mg orally, once daily for 90 days
  Arms: Rosuvastatin + Ezetimibe + Bempedoic Acid

SUMMARY:
This Open-label, randomized clinical trial evaluates the comparative efficacy and safety of dual versus triple lipid-lowering therapy using rosuvastatin, ezetimibe, and bempedoic acid in patients with type 2 diabetes mellitus and elevated LDL cholesterol. The study aims to determine whether adding bempedoic acid to standard dual therapy provides superior lipid control without compromising safety. The 126 participants, aged 35 - 60 years will be randomly assigned to one of three treatment groups for 12 weeks, and their lipid profiles, glycemic control, and adverse effects will be monitored.The total duration of study will be 6 months, with a 3 months individual treatment period.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label clinical trial conducted over a 12-week period to evaluate the comparative efficacy and safety of dual versus triple lipid-lowering therapy in patients with type 2 diabetes mellitus (T2DM) and elevated LDL cholesterol (LDL-C).

The trial includes three treatment arms, Arm A will receive Rosuvastatin + Ezetimibe, Arm B will receive Bempedoic Acid + Ezetimibe and Arm C will receive Rosuvastatin + Ezetimibe + Bempedoic Acid.

Eligible participants are adults aged 35 - 60 years with a confirmed diagnosis of type 2 diabetes mellitus and elevated LDL cholesterol despite standard care. Exclude patients with severe hepatic or renal impairment, history of gout or hyperuricemia, muscle disorders or previous statin intolerance or Participation in another clinical trial within 30 days All participants will be randomly assigned to one of the three arms. Baseline assessments include lipid profile (TC, TG, HDL, LDL, VLDL), glycemic parameters (FBS, RBS, HbA1c), creatine kinase, uric acid, and documentation of medical history and concomitant medications. Follow-up assessments will occur at week 12 to evaluate changes in primary and secondary outcomes.

The primary outcome is change in LDL cholesterol from baseline to 12 weeks and secondary Outcomes include total cholesterol (TC), high-density lipoprotein (HDL), triglycerides (TG), very-low-density lipoprotein (VLDL), creatine kinase (CK), Uric acid, glycemic control like HbA1c, fasting blood sugar (FBS), random blood sugar (RBS), safety and tolerability including muscle spasm, myalgia, or gout attacks Safety Monitoring through all adverse events will be recorded during the study. If participants reporting muscle symptoms or hyperuricemia will be evaluated promptly. Laboratory tests will be repeated at study completion or earlier if clinically indicated.

This study is designed to assess whether the addition of bempedoic acid to standard dual therapy provides superior lipid-lowering efficacy without increasing adverse events in T2DM patients with elevated LDL-C. The findings will inform clinical practice on optimal lipid-lowering strategies for high-risk diabetic patients.

The study has received approval from BUHS-IRB (#180/25) and will be conducted in accordance with Good Clinical Practice (GCP) guidelines. Written informed consent will be obtained from all participants before study procedures.

ELIGIBILITY:
Inclusion Criteria:

Males and females Age 35-60 years HbA1c ≥ 7.0 (≥ 48 mmol/mol) On stable anti-diabetic therapy for at least 3 months LDL-C > 100 mg/dL on at least two occasions Diagnosed with hypercholesterolemia Establish high cardiovascular risk (e.g, previous MI, stroke or atherosclerosis) or

* 2 cardiovascular risk factors (hypertension, smoking, obesity, family history) BMI >23 - <32(WHO Asian Criteria) No prior statin side effects

Exclusion Criteria:

HbA1c >10 % (86 mmol/mol) BMI > 32 Type 1 Diabetes, gestational diabetes Pregnancy or lactation Acute liver disease or ALT/AST levels > 3× the upper limit of normal Renal failure (GFR < 30 mL/min) Uncontrolled hypothyroidism or nephrotic syndrome Recent cancer diagnosis (last 6 months) Current use of other lipid-lowering agents (e.g., fibrates or PCSK9 inhibitors) Known allergy to any component Statin intolerance with severe adverse effects (e.g., rhabdomyolysis)

-

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Percent reduction in LDL-C and proportion of patients achieving LDL-C <70 mg/dL | 3 months
  The study will measure the percentage change in LDL-C from baseline to 12 weeks and the proportion of participants achieving LDL-C <70 mg/dL as per international guidelines to assess the efficacy of dual and triple lipid-lowering therapies in patients with Type 2 Diabetes Mellitus.

SECONDARY OUTCOMES:
Secondary outcome: Changes in Lipid Profile | 3 months
  The study will measure changes in total cholesterol, triglycerides, HDL, LDL, and VLDL from baseline to 12 weeks to evaluate the efficacy of dual and triple lipid-lowering therapies.
Secondary Outcome: Safety Monitoring by muscle and metabolic Parameters | 3 months
  The study will monitor creatine kinase and uric acid levels from baseline to 12 weeks to assess muscle-related and metabolic safety of the therapies.
Secondary Outcome : Treatment-Related Adverse Effects | 3 months
  The study will record any treatment-related adverse effects (e.g., muscle spasm, gout, gastrointestinal symptoms) over 12 weeks to assess overall safety.

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Khatoon, MBBS, Principal Investigator — Bahria University, Islamabad
Locations (1):
- National Medical Center, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) from all study participants, including demographic information, lipid profiles (TC, TG, HDL, LDL, VLDL), glycemic parameters (HbA1c, FBS, RBS), creatine kinase, uric acid, and adverse events, will be shared. Data will be fully anonymized to protect participant privacy
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available after publication of the primary study results and will remain accessible for 3 years following the study completion
Access Criteria: All data will be accessible to every one

REFERENCES:
- [Background] Laufs U, Ballantyne CM, Banach M, Bays H, Catapano AL, Duell PB, Goldberg AC, Gotto AM, Leiter LA, Ray KK, Bloedon LT, MacDougall D, Zhang Y, Mancini GBJ. Efficacy and safety of bempedoic acid in patients not receiving statins in phase 3 clinical trials. J Clin Lipidol. 2022 May-Jun;16(3):286-297. doi: 10.1016/j.jacl.2022.03.001. Epub 2022 Mar 13. PMID 35346603
- [Background] Rubino J, MacDougall DE, Sterling LR, Hanselman JC, Nicholls SJ. Combination of bempedoic acid, ezetimibe, and atorvastatin in patients with hypercholesterolemia: A randomized clinical trial. Atherosclerosis. 2021 Mar;320:122-128. doi: 10.1016/j.atherosclerosis.2020.12.023. Epub 2020 Dec 31. PMID 33514449
- [Background] Ballantyne CM, Laufs U, Ray KK, Leiter LA, Bays HE, Goldberg AC, Stroes ES, MacDougall D, Zhao X, Catapano AL. Bempedoic acid plus ezetimibe fixed-dose combination in patients with hypercholesterolemia and high CVD risk treated with maximally tolerated statin therapy. Eur J Prev Cardiol. 2020 Apr;27(6):593-603. doi: 10.1177/2047487319864671. Epub 2019 Jul 29. PMID 31357887
- [Background] Goldberg AC, Leiter LA, Stroes ESG, Baum SJ, Hanselman JC, Bloedon LT, Lalwani ND, Patel PM, Zhao X, Duell PB. Effect of Bempedoic Acid vs Placebo Added to Maximally Tolerated Statins on Low-Density Lipoprotein Cholesterol in Patients at High Risk for Cardiovascular Disease: The CLEAR Wisdom Randomized Clinical Trial. JAMA. 2019 Nov 12;322(18):1780-1788. doi: 10.1001/jama.2019.16585. PMID 31714986
- [Background] Bays HE, Banach M, Catapano AL, Duell PB, Gotto AM Jr, Laufs U, Leiter LA, Mancini GBJ, Ray KK, Bloedon LT, Sasiela WJ, Ye Z, Ballantyne CM. Bempedoic acid safety analysis: Pooled data from four phase 3 clinical trials. J Clin Lipidol. 2020 Sep-Oct;14(5):649-659.e6. doi: 10.1016/j.jacl.2020.08.009. Epub 2020 Sep 2. PMID 32980290
- [Background] Pirillo A, Catapano AL. New insights into the role of bempedoic acid and ezetimibe in the treatment of hypercholesterolemia. Curr Opin Endocrinol Diabetes Obes. 2022 Apr 1;29(2):161-166. doi: 10.1097/MED.0000000000000706. PMID 34980867
- [Background] Nissen SE, Lincoff AM, Brennan D, Ray KK, Mason D, Kastelein JJP, Thompson PD, Libby P, Cho L, Plutzky J, Bays HE, Moriarty PM, Menon V, Grobbee DE, Louie MJ, Chen CF, Li N, Bloedon L, Robinson P, Horner M, Sasiela WJ, McCluskey J, Davey D, Fajardo-Campos P, Petrovic P, Fedacko J, Zmuda W, Lukyanov Y, Nicholls SJ; CLEAR Outcomes Investigators. Bempedoic Acid and Cardiovascular Outcomes in Statin-Intolerant Patients. N Engl J Med. 2023 Apr 13;388(15):1353-1364. doi: 10.1056/NEJMoa2215024. Epub 2023 Mar 4. PMID 36876740
- [Background] Marazzi G, Caminiti G, Perrone MA, Campolongo G, Cacciotti L, Giamundo DM, Iellamo F, Severino P, Volterrani M, Rosano G. Addition of Bempedoic Acid to Statin-Ezetimibe versus Statin Titration in Patients with High Cardiovascular Risk: A Single-Centre Prospective Study. J Cardiovasc Dev Dis. 2024 Sep 14;11(9):286. doi: 10.3390/jcdd11090286. PMID 39330344
- See also: ACC/AHA cholesterol management guidelines — https://www.acc.org/latest-in-cardiology
- See also: ADA information on diabetes and cardiovascular risk. — https://www.diabetes.org/